CLINICAL TRIAL: NCT02274779
Title: Multicentric Phase II Trial of Salvage Radiotherapy Combined With Hormonotherapy in Oligometastatic Pelvic Node Relapses of Prostate Cancer (OLIGOPELVIS / GETUG P07)
Brief Title: Salvage Radiotherapy Combined With Hormonotherapy in Oligometastatic Pelvic Node Relapses of Prostate Cancer
Acronym: OLIGOPELVIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-N-2014-02
Record Dates: First submitted 2014-10-21; First posted 2014-10-24 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer,Oligometastasis,Radiotherapy,Hormonotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hight dose IMRT, ELIGARD (Experimental): * PTV1 PTV5 to 66 Gy in 30 fractions of 2.2 Gy
  * PTV Pelvis: 54 Gy in 30 fractions of 1.8 Gy
  * PTV Loge 60 Gy in 30 fractions of 2 Gy 6 Gy A complement of 3 in two additional fractions Gy may be delivered across the lodge PTV.
  * PTV Relapse Lodge: In addition to treating the PTV Lodge, additional radiation of 6 Gy in 3 fractions of 2 Gy may be made to bring the total dose of 72 Gy in 36 fractions of 2 Gy.
  Interventions: Drug: ELIGARD

INTERVENTIONS:
Drug: ELIGARD — Hormone therapy is recommended Eligard 45 mg acting for 6 months. It will be ideally administered the day of start of radiation therapy or within 3 months before the first day of radiotherapy.
  Nevertheless, free prescription is left to investigators. When using other hormonal strategies (anti-androgen agonists, LHRH antagonists or LHRH), an administration for six months will be critical.
  Other Names: Leuproréline

SUMMARY:
There is an increasing number of reports describing the existence of a proportion of prostate cancer patients who present with a reduced number of metastases (<5 lesions) at relapse. This oligometastatic status has also been recognized in other tumor types such as melanoma, soft tissue sarcoma, liver, lung, and breast cancer, and has influenced the management of these malignancies in that a more radical treatment such as surgical resection has been employed. Positron Emission Tomography-Computed Tomography (PET-CT) studies with tracers such as choline or acetate are reliable tools to help with the diagnosis of oligometastatic disease after biochemical treatment failure in prostate cancer. An aggressive treatment combining androgen depriving therapy (ADT) and and high-dose irradiation to the oligometastatic lesions, as detected by PET-CT, may be proposed for these oligometastatic patients. Such a treatment strategy may hypothetically succeed to prolong the failure-free interval between two consecutive ADT courses, or even cure selected patients with limited metastatic burden. In this study the investigators plan to assess biochemical or clinical relapse-free survival at 2 years of prostate cancer with 1-5 oligometastases treated concomitantly with high-dose conformal Radiation Therapy and LH-RH agonists.

DETAILED DESCRIPTION:
1. Hormonotherapy

   Hormone therapy is recommended Eligard 45 mg acting for 6 months. It will be ideally administered the day of start of radiation therapy or within 3 months before the first day of radiotherapy.

   Nevertheless, free prescription is left to investigators. When using other hormonal strategies (anti-androgen agonists, LHRH antagonists or LHRH), an administration for six months will be critical.
2. Radiotherapy

Conformational Radiotherapy techniques in Intensity-Modulated (IMRT)

2.1) Doses prescribed

* PTV1 PTV5 to 66 Gy in 30 fractions of 2.2 Gy
* PTV Pelvis: 54 Gy in 30 fractions of 1.8 Gy
* PTV Loge 60 Gy in 30 fractions of 2 Gy 6 Gy A complement of 3 in two additional fractions Gy may be delivered across the lodge PTV.
* PTV Relapse Lodge: In addition to treating the PTV Lodge, additional radiation of 6 Gy in 3 fractions of 2 Gy may be made to bring the total dose of 72 Gy in 36 fractions of 2 Gy.

2.2) Treatment

Radiation Guided by a picture (IGRT) will be performed daily. This daily recalibration will be based at least on bone structures. It will be possible to readjust the nodal structures.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven adenocarcinoma of the prostate
2. Patients aged 18 years or more
3. PS 0-1
4. Previous radical treatment to the prostate (radiotherapy or surgery)
5. PSA increase of at least 3 assays in the same laboratory over the last 12 months.
6. 1-5 pelvic lymph node metastases detected with 18FCH-PET. A relapse in the dressing prostatectomy is associated possible.
7. Upper limit of lymph node metastases: aortic bifurcation
8. Respect dosimetric constraints to organs at risk
9. Treatment with hormone therapy may be started before inclusion, to a maximum of three months prior to Day 1 of radiotherapy. This hormone will necessarily be preceded by a free interval treatment of at least 6 months since the last injection, by adding the duration of action of this predictable injection (1, 3 or 6 months)
10. Patient affiliated to a social security scheme
11. Patient Information and written informed consent form signed

Exclusion Criteria:

1. bone or visceral metastatic relapse associated
2. para-aortic nodal relapse (the upper limit is tolerated aortic bifurcation)
3. more than 5 lymph node metastases
4. Proof of metastases at initial diagnosis
5. Evidence of distant metastases in the pelvic lymph nodes or outside the prostate bed
6. prior pelvic lymph nodes Irradiation. Irradiation of the bed of the prostate is not an exclusion criterion, but the junction between prior irradiation bed prostatectomy and radiation field pelvic lymph nodes should be examined carefully
7. castration resistance defined by clinical or biochemical progression despite a combined androgen blockade
8. known contraindications to pelvic irradiation (eg, chronic inflammatory bowel disease, ...)
9. known contraindications to hormone therapy, according to standard recommendations in force
10. serious Hypertension not controlled by appropriate treatment
11. Other concomitant cancer or history of cancer (within 5 years prior to study entry), except basal cell or squamous cell carcinomas of the skin.
12. Patient with a psychological, familial, sociological or geographical potentially hampering compliance with the study protocol and follow-up schedule
13. Patient already included in another interventional study involving the approval of a CPP during his screening for the study OLIGOPELVIS
14. Private person of liberty or major trust

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
biochemical or clinical relapse-free survival at 2 years | 2 years
  The biochemical or clinical relapse is defined by:
  * a PSA level greater than the PSA before treatment, with two successive elevations in the same laboratory
  * and / or an increase in the number of metastatic sites at the evaluation visit

SECONDARY OUTCOMES:
gastrointestinal toxicities after radiation | 1 month (acute toxicities) and 2 years (late toxicities)
  main toxicities expected are : proctitis, ileitis, diarrhea
Local relapse versus distant relapse | expected up to 24 month
  Medical imaging exams will be performed every 6 month for 2 years, and then every years until patient progression
Overall survival | every year
  overall survival will be assessed every year during patient life

CONTACTS AND LOCATIONS:
Overall Officials: SUPIOT Stéphane, MD, Principal Investigator — Institut de Cancérologie de l'Ouest (ICO) - Nantes, France
Locations (2):
- France (2):
  - ICO Paul Papin, Angers
  - ICO René Gauducheau, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Supiot S, Rio E, Pacteau V, Mauboussin MH, Campion L, Pein F. OLIGOPELVIS - GETUG P07: a multicentre phase II trial of combined salvage radiotherapy and hormone therapy in oligometastatic pelvic node relapses of prostate cancer. BMC Cancer. 2015 Sep 25;15:646. doi: 10.1186/s12885-015-1579-0. PMID 26408012
- [Derived] Ploussard G, Almeras C, Briganti A, Giannarini G, Hennequin C, Ost P, Renard-Penna R, Salin A, Lebret T, Villers A, Soulie M, de la Taille A, Flamand V. Management of Node Only Recurrence after Primary Local Treatment for Prostate Cancer: A Systematic Review of the Literature. J Urol. 2015 Oct;194(4):983-8. doi: 10.1016/j.juro.2015.04.103. Epub 2015 May 9. PMID 25963190